CLINICAL TRIAL: NCT00016016
Title: A Phase I/II Study of Flavopiridol (NSC 649890, IND 46,211) in Timed Sequential Combination With Cytosine Arabinoside (Ara-C) and Mitoxantrone for Adults With Poor-Risk Acute Leukemias
Brief Title: Flavopiridol, Cytarabine, and Mitoxantrone in Treating Patients With Acute Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03153; NCI-2012-03153 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSGCC-0052; NCI-3170; JHOC-J0254; J0254 (Other: Johns Hopkins University); 3170 (Other: CTEP); U01CA070095 (NIH); U01CA069854 (NIH)
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Cytarabine; Mitoxantrone; alvocidib

ARMS (1):
- Treatment (flavopiridol, cytarabine, mitoxantrone) (Experimental): Patients receive flavopiridol IV over 1 hour on days 1-3 and cytarabine IV continuously on days 6-9 followed by mitoxantrone IV over 30-150 minutes on day 9. Patients achieving a partial or complete response after the first course of therapy may receive an additional course of therapy beginning 35 ± 7 days after blood count recovery.
  Interventions: Drug: cytarabine; Drug: mitoxantrone hydrochloride; Drug: alvocidib; Other: pharmacological study; Other: laboratory procedure

INTERVENTIONS:
Drug: cytarabine — Given IV
Drug: mitoxantrone hydrochloride — Given IV
Drug: alvocidib — Given IV
Other: pharmacological study — Correlative studies
Other: laboratory procedure — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining flavopiridol and cytarabine with mitoxantrone in treating patients who have acute leukemia. Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities of escalating doses of flavopiridol administered in a timed sequence with ara-C and mitoxantrone in adults with refractory or relapsed acute leukemias or high-risk myelodysplasias (MDS).

II. To determine if flavopiridol administered in a timed sequence with ara-C and Mitoxantrone will induce clinical responses in adults with refractory or relapsed acute leukemias or MDS.

III. To determine if flavopiridol is directly cytotoxic to leukemic blasts in vivo.

IV. To determine if flavopiridol can recruit and synchronize residual leukemic blasts to proliferate in vivo.

OUTLINE: This is a dose-escalation study of flavopiridol. (Phase I closed to accrual effective10/24/2003).

Patients receive flavopiridol IV over 1 hour on days 1-3 and cytarabine IV continuously on days 6-9 followed by mitoxantrone IV over 30-150 minutes on day 9. Patients achieving a partial or complete response after the first course of therapy may receive an additional course of therapy beginning 35 ± 7 days after blood count recovery.

Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. (Phase I closed to accrual effective 10/24/2003). Once the MTD is reached, additional patients are accrued to receive flavopiridol at the recommended phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnoses of poor-risk hematologic malignancies will be considered eligible for this Phase I/II study
* Pathological confirmation of the diagnosis of AML or ALL
* ECOG performance status 0,1,2
* Patients must be able to give informed consent
* Female patients of childbearing age must have negative pregnancy test
* AST and ALT =< 2.5 x normal
* Alkaline phosphatase =< 2.5 x normal
* Bilirubin =< 1.5 x normal
* Serum creatinine =< 2.0 mg/dl
* Left ventricular ejection fraction must >= 45% by MUGA or Echocardiogram
* Acute Myelogenous Leukemia (AML)

  * AML arising from MDS
  * Secondary AML
  * Relapsed or refractory AML, including primary induction failure
* Acute Lymphoblastic Leukemia (ALL)

  * Relapsed or refractory ALL, including primary induction failure
  * Patients who fail primary induction therapy or who relapse after achieving complete remission (CR) are eligible if they have undergone no more than 3 prior courses of induction/reinduction
* There should be an interval of at least 4 weeks from any previous intensive chemotherapy before beginning flavopiridol, with the exceptions non-aplasia producing treatments (i.e. hydroxyurea, interferon, imatinib, 6MP, thalidomide); patients should have recovered completely from any treatment-related toxicities; patients may have received hematopoietic growth factors previously, but must be off all growth factors (including EPO, G-CSF, GM-CSF, IL-3, IL-11) for at least 4 days prior to beginning flavopiridol
* Patients who have undergone stem cell transplantation (SCT), autologous or allogeneic, are eligible provided that they are >= 4 weeks from stem cell infusion, have no active GVHD, and meet other eligibility criteria

Exclusion Criteria:

* Hyperleukocytosis with >= 50,000 leukemic blasts/mm^3
* Active, uncontrolled infection
* Disseminated intravascular coagulation
* Active CNS leukemia
* Concomitant chemotherapy, radiation therapy or immunotherapy
* Intrinsic impaired cardiac function (MI within the preceding 3 months or history of severe coronary artery disease, cardiomyopathy, CHF > Class II)
* History of congestive heart disease, or arrhythmia without regard to time, severity or resolution
* Women who are pregnant or lactating will not be eligible for this trial, as the investigational agent may be harmful to the developing fetus or nursing infant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2001-02; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) as assessed by NCI CTC version 2.0 | Up to 35 days
Complete remission (CR) | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Judith Karp, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States